CLINICAL TRIAL: NCT03220347
Title: A Phase 1, Open-label, Dose-finding Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of CC-90010 in Subjects With Advanced Solid Tumors and Relapsed/Refractory Non-Hodgkin's Lymphomas
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of CC-90010 in Subjects With Advanced Solid Tumors and Relapsed/Refractory Non-Hodgkin's Lymphomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-90010-ST-001; U1111-1194-8570 (Registry Identifier: WHO); 2015-004371-79 (EudraCT Number)
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Lymphoma, Non-Hodgkin; Neoplasms
Keywords: Non-Hodgkin's Lymphomas; Safety; Efficacy; CC-90010; Solid Tumors; Relapsed/Refractory
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CC-90010 in patients with solid tumors and NHL (Experimental): Subjects will be administered orally once daily for 3 consecutive days followed by 4 consecutive days off drug every week (3/7-days schedule) in each 28 day cycle in Part A. Alternative dosing schedules (eg, 2-days-on/5-days- off each week, 3-days-on/4-days-off every other week, 4-days on/24 days off) may be evaluated one dosing schedule at a time or ≥ 2 dosing schedules given in parallel, based on the review of available safety, PK, pharmacodynamic (PD), and efficacy data.
  Interventions: Drug: CC-90010

INTERVENTIONS:
Drug: CC-90010 — CC-90010 is an oral, potent and reversible inhibitor of the epigenetic target bromodomain and extra-terminal (BET) proteins.

SUMMARY:
Study CC-90010-ST-001 is an open-label, Phase 1a, dose escalation and expansion, First-in-human (FIH) clinical study of CC-90010 in subjects with advanced or unresectable solid tumors and relapsed and/or refractory advanced Non-Hodgkin's lymphoma (NHL). The dose escalation part (Part A) of the study will explore escalating oral doses of CC-90010 to estimate the maximum tolerated dose (MTD) of CC-90010. The expansion part (Part B) will further evaluate the safety and efficacy of CC-90010 administered at or below the MTD in the following cohorts:

Cohort 1: relapsed and/or refractory DLBCL approximately 20-25 evaluable subjects at 45 mg CC-90010 4-days-on/24-days-off in each 28-day cycle Cohort 2: advanced BCC -enrollment stopped due to recruitment challenges Cohort 3: relapsed and/or refractory DLBCL -approximately 15 evaluable subjects at 30mg CC-90010 3-dayson/11-days-offin each 28-day cycle.

The enrollment of subjects with R/R DLBCL in Cohort 1 and Cohort 3 was closed due to Company's strategic decision and not due to any safety concern or lack of preliminary antitumor efficacy.

The food effect assessment (Part C, Spain only) will evaluate the impact of food on CC-90010 when administered at the RP2D of 45 mg 4-days-on/24-days-off (180 mg per 28-day cycle), by comparison of the PK parameters following fasted and fed (high-fat, high-calorie meal) conditions.

DETAILED DESCRIPTION:
Parts A, B and C will consist of 3 periods: Screening, Treatment and Follow-up.

Screening Period:

The Screening Period starts 28 days (± 3 days) prior to first dose of CC-90010. The informed document (ICD) must be signed and dated by the subject and the administering staff prior to the start of any other study procedures. All screening tests and procedures must be completed within the 28 days (±3 days) prior to the first dose of CC-90010.

Treatment Period:

During the Treatment Period, CC-90010 was initially administered orally once daily for 3 consecutive days followed by 4 consecutive days off drug every week (3/7-days schedule) in each 28-day cycle in Part A. Alternative dosing schedules (eg, 2-days-on/5-days- off each week, 3-days-on/4-days-off every other week, 4-days on/24 days off) may be evaluated one dosing schedule at a time or ≥ 2 dosing schedules given in parallel, based on the review of available safety, PK, pharmacodynamic (PD), and efficacy data by the SRC.

Following completion of dose escalation in Part A, selected expansion cohorts will receive CC-90010 in Part B. The SRC determined the RP2D for Part B to be 45 mg CC-90010 given once daily for 4 consecutive days on followed by 24 consecutive days off (4-days-on/24-days-off) in each 28-day cycle. There are 3 cohorts in Part B expansion. A cohort of up to approximately 20-25 subjects with relapsed and/or refractory DLBCL (Cohort 1) enrolled at the RP2D..

Enrollment in advanced BCC (Cohort 2) will be stopped due to recruitment challenges. An additional cohort of approximately 15 evaluable subjects with R/R DLBCL (Cohort 3) will be enrolled under an alternative dosing regimen of 30 mg CC-90010 3days-on/11-days off in each 28-day cycle. The enrollment of subjects with R/R DLBCL in Cohort 1 and Cohort 3 was closed due to Company's strategic decision and not due to any safety concern or lack of preliminary antitumor efficacy. The food effect assessment (Part C, Spain only) will evaluate the impact of food on CC-90010 when administered at the RP2D of 45 mg 4-days-on/24-days-off, by comparison of PK parameters following fasted and fed (high-fat, high-calorie meal) conditions in approximately 24 subjects with advanced solid tumors.

Follow-up Period:

In the Follow-up Period, subjects will be followed for 28 days (± 3 days) after the last dose of CC-90010 for safety.

After the Safety Follow-up visit, all subjects will be followed every subsequent 3 months (± 2 weeks) for survival follow-up for up until 2 years or until death, lost to follow-up, or the End of Trial, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Age = or > 18 years.
2. For subjects enrolling in food-effect assessment (Part C) only: a. Subject must agree and be willing to consume a standard high-fat, high-calorie meal. b. Subject must be willing to refrain from caffeine or xanthene-containing products (coffee, tea, cola, chocolate, etc.) for 48 hours prior to dosing on Cycle 1 Day 4 and Cycle 2 Day 4 and up to 24 hours post dose.
3. Subjects with histological or cytological confirmation of either:

   1. In Part A, advanced or unresectable solid tumors or advanced relapsed and/or refractory Non-Hodgkin lymphoma (ie, Diffuse large B-cell lymphoma and Follicular lymphoma or Marginal zone lymphoma) including those who have progressed on (or not been able to tolerate due to medical comorbidities or unacceptable toxicity) standard anticancer therapy or for whom no other approved conventional therapy exists.
   2. In Part B dose expansion, - Cohorts 1 and 3: relapsed and/or refractory DLBCL following at least 2 prior lines of therapy (e.g. have failed at least one line of standard therapy and have received at least one prior line of salvage therapy) OR have failed at least one prior line of standard therapy and are not eligible for autologous stem cell transplant (ASCT) or have declined ASCT; transformed lymphoma following chemotherapy for lower grade lymphoma and at least two standard treatment regimen for DLBCL.

      Subjects with two or more lines of systemic therapy must have been treated with and have lack of response after chimeric antigen receptor (CAR) T-cell therapy, if such therapy is available, OR be ineligible for CAR T-cell therapy at the time of enrollment, OR subject declined CAR T-cell therapy.

      - Cohort 2: advanced basal cell carcinoma including those who have progressed on (or not been able to tolerate due to medicalcomorbidities or unacceptable toxicity) standard anticancer therapy or for whom no other approved conventional therapy exists.

      In Part C, advanced or unresectable solid tumors including those who have progressed on (or not been able to tolerate due to medical comorbidities or unacceptable toxicity) standard anticancer therapy or for whom no other approved conventional therapy exist
4. At least one site of measurable disease for subjects with solid tumors; bi-dimensionally measurable disease on cross sectional imaging with at least one lesion >1.5 cm for subjects with NHL. For subjects with rare malignancies evaluable disease can be considered.
5. Tumor biopsies whenever safe and feasible will be collected in Part A, except for subjects with GBM. Subject consents to mandatory tumor biopsies (Screening and on treatment) in Part B. In exceptional circumstances an exemption waiver may be granted by the Sponsor for this criterion
6. ECOG PS of 0 to 1.
7. Females of childbearing potential (FCBP)1 must:

   • Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with, at least two effective contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner), one of which must be barrier, from signing the ICD, throughout the study (including dose interruptions), and for up to 6 months and 16 days following the last dose of CC-90010; and
   * Avoid conceiving for 6 months and 16 days after the last dose of CC-0010.
   * Agree to not donate oocytes while receiving CC-90010 and for 6 months and 16 days after the last dose of CC-90010.
8. Males must practice true abstinence2 (which must be reviewed on a monthly basis) or agree to use a condom (a latex condom is recommended) during sexual contact with a pregnant female or a FCBP and will avoid conceiving from signing the ICD, while participating in the study, during dose interruptions, and for at least 106 days following CC-90010 discontinuation, even if he has undergone a successful vasectomy. Additionally, subjects must not donate sperm during this same time period.

Exclusion Criteria:

Principal Exclusion Criteria

1. Subject has received anti-cancer therapy (either approved or investigational) within <or= 4 weeks or 5 half-lives, whichever is shorter prior to starting CC-90010.
2. Subject has received prior CAR T-cell therapy or other T-cell targeting treatment (approved or investigational) ≤ 4 weeks prior to starting CC-90010.
3. Toxicities resulting from prior systemic cancer therapies must have resolved. to ≤ NCI CTCAE Grade 1 prior to starting CC-90010 treatment
4. Subject has received autologous hematologic stem cell transplant (HSCT) <or= 3 months prior to starting CC-90010 treatment. Subjects with allogeneic HSCT will not be allowed on this protocol.
5. Major surgery <or= 4 weeks or minor surgery <or= 2 weeks prior to starting CC-90010 or subjects who have not recovered from surgery.
6. Completed radiation treatment < 4 weeks prior to starting CC-90010.
7. Symptomatic, untreated, or unstable central nervous system (CNS) metastases.
8. Known symptomatic acute or chronic pancreatitis.
9. Impaired cardiac function or clinically significant cardiac diseases.
10. Pregnant or nursing females.

12. History of concurrent second cancers requiring active, ongoing systemic treatment.

13. History of clinically significant cognitive disorder(s) or active cognitive disorder(s).

13. Evidence of history of bleeding diathesis. 14. Subjects with known prior episodes of non-arteritic anterior ischemic optic neuropathy (NAION) should be excluded from the study. CC-90010 should be used with caution in subjects with retinitis pigmentosa 15. Any significant medical condition that would prevent the subject from participating (or compromise compliance) in the study or would place the subject at unacceptable risk if he/she were to participate in the study.

16. Patients with poor bone marrow reserve as assessed by the Investigator such as in the following conditions:

* Having received extensive bone radiotherapy
* Having experienced several episodes of bone marrow aplasia in previous treatments
* Confirmed histological bone marrow cancer infiltration (with exemption of NHL)
* Requiring regular hematopoietic support (blood transfusion, erythropoietin, GCSF) 17. Previous SARS-CoV-2 infection within 10 days for mild or asymptomatic infections or 20 days for severe/critical illness prior to C1D1

  * Acute symptoms must have resolved and based on investigator assessment in consultation with the medical monitor, there are no sequelae that would place the subject at a higher risk of receiving study treatment.

    18. Previous SARS-CoV-2 vaccine within 7 days of C1D1. For vaccines requiring more than one dose, the full series (e.g. both doses of a two-dose series) should be completed prior to C1D1 when feasible and when a delay in C1D1 would not put the study subject at risk.
  * The administration of a live SARS-CoV-2 vaccine is prohibited up to 14 days prior to the initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to 7 years
  Number of participants with adverse events
Dose Limiting Toxicities (DLTs) | Up to 7 years
  A DLT is defined as any of the toxicities described in the protocol occurring within the DLT assessment unless the event can clearly be determined to be unrelated to CC-90010
Maximum tolerated dose (MTD) | Up to 7 years
  The MTD is the highest dose that causes DLTs in not more than 33% of the subjects treated with CC-90010 in the first cycle with at least 6 evaluable subjects treated at this dose.

SECONDARY OUTCOMES:
Clinical benefit rate (CBR) | Up to 7 years
  Is defined as tumor responses (as assessed by the Investigators) of complete response (CR), partial response (PR) and stable disease (SD) (SD of ≥ 4 months duration).
Objective response rate (ORR) | Up to 7 years
  Is defined as the percent of subjects whose best response is CR or PR.
Duration of Response Rate | Up to 7 years
  Is measured from the time when criteria for CR/PR are first met (whichever is first recorded) until the first date at which progressive disease is objectively documented
Duration of stable disease | Up to 7 years
  For subjects with best response of SD, duration of SD is measured from the first dose date until the criteria for progression are met
Progression-free survival (PFS) | Up to 7 years
  Is defined as the time from the first dose of CC-90010 to the first occurrence of disease progression or death from any cause.
Overall survival | Up to 7 years
  Is measured as the time from the first dose of CC-90010 to death due to any cause.
Pharmacokinetic- Cmax | Up to 7 years
  Maximum observed plasma concentration on first and last day of dosing within a cycle
Pharmacokinetic- AUC | Up to 7 years
  Area under the plasma concentration time-curve on first and last day of dosing within a cycle
Pharmacokinetic- Tmax | Up to 7 years
  Time to maximum plasma concentration on first and last day of dosing within a cycle
Pharmacokinetic- t1/2 | Up to 7 years
  Terminal half-life on last day of dosing within a cycle
Apparent Clearance | Up to 7 years
  Apparent total systemic clearance to be estimated following the last dose in cycle 1
Apparent Volume of Distribution | Up to 7 years
  Apparent steady state volume of distribution to be estimated following the last dose in cycle 1
Pharmacokinetic- AUClast | Up to 7 years
  Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration
Pharmacokinetic- AUC0-24 | Up to 7 years
  Area under the plasma concentration-time curve calculated from time zero to 24 hours
Pharmacokinetic- AUC0-∞ | Up to 7 years
  Area under the concentration-time curve calculated from time zero to infinity

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (11):
- France (2):
  - Local Institution - 102, Bordeaux
  - Local Institution - 100, Villejuif
- Italy (3):
  - Local Institution - 303, Meldola
  - Local Institution - 301, Napoli, Campania
  - Local Institution - 302, Rozzano (MI)
- Japan (3):
  - Local Institution - 400, Kashiwa-shi, Chiba
  - Local Institution - 402, Koto-ku, Tokyo
  - Local Institution - 401, Chikusa-ku
- Spain (3):
  - Local Institution - 200, Barcelona
  - Local Institution - 201, Madrid
  - Local Institution - 202, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com